CLINICAL TRIAL: NCT06013384
Title: Clinical Feasibility of Low Intensity Focused Ultrasound Pulsation for the Treatment of Treatment Resistant Major Depressive Disorder
Brief Title: Low-Intensity Focused Ultrasound for Treatment-Resistant Depression
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study PI left institution and there is currently no one else available to run the study.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00128763
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
Keywords: focused ultrasound; neuromodulation
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active/Active Group (Experimental): This group will receive eight total treatments of LIFUP across two days one week apart (four treatments each day).
  Interventions: Device: Low-Intensity Focused Ultrasound Pulsation
- Sham/Active Group (Other): This group will receive sham LIFUP for four treatments over one day, followed by four total treatments of active LIFUP across one day one week after sham.
  Interventions: Device: Low-Intensity Focused Ultrasound Pulsation; Device: Sham Low-Intensity Focused Ultrasound Pulsation

INTERVENTIONS:
Device: Low-Intensity Focused Ultrasound Pulsation — Low-intensity focused ultrasound pulsation will be directed towards the target region at FDA-approved intensity levels in treatment sessions one and two.
Device: Sham Low-Intensity Focused Ultrasound Pulsation — Sham low-intensity focused ultrasound pulsation will be given.
  Arms: Sham/Active Group

SUMMARY:
The Investigators are proposing to demonstrate safety and efficacy of LIFUP for treatment resistant major depressive disorder in a ten-patient pilot study. LIFUP is an emerging treatment with the advantage of being able to target subcortical transcranial targets, which may have superior efficacy or a shorter treatment course compared to other available treatments such as transcranial magnetic stimulation. This study will investigate the effect of this stimulation on the left subgenual cingulate cortex, a highly connected node in the depression network that is correlated with clinical symptomatology.

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate safety and efficacy of a novel treatment, low intensity focused ultrasound pulsation (LIFUP) for treatment resistant depression (TRD). Participants will receive either LIFUP or sham stimulation with crossover of sham participants into the treatment group halfway through the treatment course. The initial visit will involve consent and an MRI scan, followed by several more either active or sham treatments outside of the MRI environment delivered over the course of two days over one week. Response and potential side effects will be monitored pre- and post- each treatment along with one week and one month follow-up assessments.

ELIGIBILITY:
Inclusion criteria:

* Male or female
* Age 18-70
* Normal or corrected-to normal vision and hearing
* Primary diagnosis of major depressive disorder, moderate/severe per DSM-5 (MADRS >20)
* The duration of the illness must exceed one year
* Must be medically stable as determined by investigator
* Patient must have attempted and failed treatment with at least 2 SSRI and 1 augmentation
* History of rTMS is permitted, but not required

Exclusionary criteria:

* Diagnosis of primary DSM-5 depressive disorder other than MDD
* Anxiety disorders such as GAD are permitted as long as MDD is primary
* Diagnosis of schizophrenia or bipolar disorder
* Current use of any non-prescribed psychoactive medications or drugs (aside from medications for treatment of MDD)
* Contraindication to enter the MRI environment.
* Pregnancy (or suspected/possible pregnancy or plan to become pregnant in the short term).
* Urine Pregnancy Test: If the subject is a woman of childbearing potential and /or a man capable of fathering a child before, during, and/or after participation precaution should be taken. Examples of acceptable methods of birth control for participants involved in the study includes: birth control pills, patch, IUD, condom, sponge, diaphragm with spermicide, or avoiding sexual activity that could cause the subject to become pregnant.
* Inability to adhere to treatment schedule.
* Initiation of new antidepressant treatment at the time of study randomization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) Score Change | One week post-treatment
  Change in the MADRS score, which ranges from 0-60, with 0-8 = no depression; 9-17 = mild; 18-34 = moderate; and >35 = severe

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) Score Change | One week post-treatment
  Change in PHQ-9 Score, which ranges from 0-27, with 0-4 = no depression; 5-9 = mild; 10-14 = moderate; and >15 = severe
General Anxiety Disorder (GAD-7) Score Change | One week post-treatment
  Change in GAD-7 Score, which ranges from 0-21, with 0-4 = no anxiety; 5-9 = mild; 10-14 = moderate; and >15 = severe

CONTACTS AND LOCATIONS:
Locations (1):
- 30 Bee Street, Charleston, South Carolina, United States